CLINICAL TRIAL: NCT03180281
Title: Exploring Effective and Safety Therapies Which Protect Islet β Cell on Newly Diagnosed Type 2 Diabetes Patients With High Glucose Toxicity
Brief Title: Therapies on Newly Diagnosed Type 2 Diabetes Patients With High Glucose Toxicity Which Protect Islet β Cell
Acronym: TOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2016LSL-048
Record Dates: First submitted 2017-03-20; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Insulin; Insulin Glargine; Insulin Detemir; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DPP4 group (Experimental): DPP4 inhibitor,1 pill qd
  Interventions: Drug: DPP4
- insulin group (Experimental): insulin,glargine or detemir，0.2U/Kg,qd
  Interventions: Drug: Insulin
- SU group (Placebo Comparator): SU,Glimepiride，1-2mg qd
  Interventions: Drug: SU

INTERVENTIONS:
Drug: DPP4 — sitagliptin phosphate 100mg qd
  Other Names: sitagliptin phosphate
  Arms: DPP4 group
Drug: Insulin — Insulin Glargine or detemir 0.2U/kg qd
  Other Names: Glargine or detemir
  Arms: insulin group
Drug: SU — Glimepiride 1-2mg qd
  Other Names: Glimepiride
  Arms: SU group

SUMMARY:
Prevalence of diabetes is increasing rapidly both in China and all over the world.Hyperglycemia is an important risk factor and major hazard to cardiovascular and cerebrovascular diseases and even dangerous to human health."High glucose toxicity "cause pancreatic β cell non-physiologic and irreversible damage.It is an important cause of β cell dysfunction.High glucose toxicity further suppresses insulin secretion of β cell, further even β-cell function failure.It is urgent to explore more effective and safety treatments which can also protect islet cells function.How to release high glucose toxicity , reverse the toxic effects of hyperglycemia on islet β cells as early as possible, and to maximize recover and protect the pancreatic β cell function is the keypoints of this study.Our aim is to explore the non-inferiority of new antidiabetic drugs DPP4 inhibitors on releasing glucose toxicity and protecting islet β cell function compared with traditional treatments on newly diagnosed type 2 diabetes,compare efficacy and safety of different oral antidiabetic drugs and insulin on newly diagnosed type 2 diabetes patients with high glucose toxicity and compare differences of different oral antidiabetic drugs and insulin on protecting pancreatic β-cell function.

DETAILED DESCRIPTION:
Patients were divided into 3 groups:

1. DPP-4 inhibitor treatment group (45 cases): DPP-4 inhibitor (sitagliptin phosphate) combined with metformin and/or acarbose;
2. insulin treatment group (45 cases): insulin (insulin glargine or insulin detemir) and/or metformin;
3. Sulfonylureas treatment group (45 cases): sulfonylureas combined with metformin and/or acarbose;

ELIGIBILITY:
Inclusion Criteria:

* newly onset
* type 2 diabetes
* BMI 18-30kg/m2
* FBS≧11.1mmol/L，GHbA1c≧9%
* urine ket ≦(1+)
* Normal liver and kidney function

Exclusion Criteria:

* type 1 diabetes
* renal or hepatic insufficiency
* Severe ketoacidosis
* Treatment with corticosteroids, immunosuppressive agents or cytotoxic drugs
* Severe systemic disease
* History of pancreatitis or pancreatic surgery
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose,glycosylated hemoglobin(GHbA1c) | From date of randomization until the date of first documented progression, assessed up to 3 months
  mmol/L,%

SECONDARY OUTCOMES:
weight loss | From date of randomization until the date of first documented progression, assessed up to 3 months
  kilograms
Lipid changes | From date of randomization until the date of first documented progression, assessed up to 3 months
  mmol/L
Incidence of hypoglycemia | From date of randomization until the date of first documented progression, assessed up to 3 months
  times

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sui, Doctor, Principal Investigator — First Affiliated Hospital of Xi'an Jiao Tong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He M, Deng M, Wang J, Fan P, Wang Y, Zhao X, He Y, Shi B, Sui J. Efficacy and tolerability of sitagliptin and metformin compared with insulin as an initial therapy for newly diagnosed diabetic patients with severe hyperglycaemia. Exp Ther Med. 2021 Mar;21(3):217. doi: 10.3892/etm.2021.9649. Epub 2021 Jan 15. PMID 33574913